CLINICAL TRIAL: NCT04370002
Title: Leveraging Artificial Intelligence for the Assessment of Severity of Depressive Symptoms
Brief Title: Sensor-based Characterization of Depression
Acronym: SENSCODE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Paola Pedrelli, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2019P000997
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Unipolar Depression
Keywords: Depression; Sensors
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: This is an observational study. There is no active treatment that is examined.

SUMMARY:
This is a longitudinal study where individual with Major Depressive Disorder (MDD) will be monitored for 12 weeks. The study aims to develop an objective, sensor-based, algorithm able to detect the presence of depression as well as predict treatment response. Measurement-based treatment is considered optimal and the development of a valid passive, objective, behavioral and biological assessment of depressive symptoms that does not rely on clinician interviews will improve monitoring and ultimately improve treatment significantly.

DETAILED DESCRIPTION:
In this longitudinal study 100 individuals with Major Depressive Disorder (MDD) will be monitored for 12 weeks. Data will include self-report surveys, in-person assessments, physiological features derived by wearable devices and socialization and activity data derived by mobile applications. The study will utilize advanced statistical methods to integrate different sources of passive sensor-based behavioral and physiological data to develop models able to detect depression and predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (ages 18-75),
2. Able to read, understand, and provide written informed consent in English,
3. Meet criteria for a primary psychiatric diagnosis of current major depressive disorder
4. Hamilton Depression Rating Scale (HDRS) total score ≥ 18,
5. Must have measurable skin conductance/electrodermal activity (as assessed at the screening visit),
6. Must own a working smartphone and use it regularly,
7. Must own a windows PC (or tablet) or a Mac computer (or laptop),
8. Must have access to Internet service every day.
9. Must have started antidepressant medications, changed medication dosage, or started therapy within 3 weeks

Exclusion Criteria:

1. Active drug or alcohol use disorder in the past 3 months,
2. History of psychotic disorder,
3. History of mania or hypomania,
4. Epilepsy or history of Seizure Disorder (including PNES), narcolepsy, Alzheimer Disease, Parkinson's Disease, ALS, Severe TBI, Dementia, MS, Cerebral Palsy, and Neuralgia.
5. Untreated hypothyroidism,
6. Unstable medical disease,
7. Cognitive impairment that would impede adherence to study procedures,
8. Acute suicide or homicide risk,
9. Current treatment with electroconvulsive therapy, vagal nerve stimulation therapy, deep brain stimulation, transcranial magnetic stimulation therapy, or phototherapy,
10. Cannot comprehend or communicate in English,
11. Lack of working smartphone or lack of daily access to Internet service,
12. Inability to measure skin conductance/electrodermal activity (as assessed at the screening visit), and
13. Inability or unwilling to, at minimum, wear the physiological sensor (E4) wristbands, download monitoring apps, and fill out the surveys.
14. Participants with more than two treatment failures (more than two adequate trials of meds on the basis of ATRQ) in the current mood episode.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be individuals with Major Depressive Disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale (HDRS) 17-items | Past week.
  The HDRS-17 is a clinician-based assessment of depressive symptoms. Higher scores indicate worse symptoms. Total score can range from 0 to 53.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Past 7 days
  The PHQ-9 is a self-report questionnaire of depressive symptoms. Total scores can vary from 0 to 27. Higher scores indicate worse depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Depression Clinical Research Program, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided